CLINICAL TRIAL: NCT01658358
Title: A Phase I/II Study of Lapatinib (Tykerb) Plus Liposomal Doxorubicin Hydrochloride ( Lipo-Dox) for Patients With ErbB2 Positive Metastatic Breast Cancer
Brief Title: ErbB2 Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Fang Chiu, Vice Superintendent, Cancer Center, China Medical University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF114081
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Breast Cancer
Keywords: ErbB receptor; tyrosine kinase inhibitor; Anthracycline
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I part :Systemic Therapy (Experimental): * Drug: Lapatinib
  * Drug: Lipo-Dox
  Interventions: Drug: Lapatinib; Drug: Lipo-Dox
- Phase II part (Experimental): * Drug: Lapatinib
  * Drug: Lipo-Dox Patients will receive recommended dose according to phase I study result. at least 8 cycles, then, with continue combination treatment cycles or single lapatinib treatment (start with 1500 mg per day) at investigator's discretion.
  Interventions: Drug: Lapatinib; Drug: Lipo-Dox

INTERVENTIONS:
Drug: Lapatinib — * dose level I, II 1000mg po daily
  * dose level III, IV 1250mg po daily
  Other Names: Tykerb
Drug: Lipo-Dox — at the dose level reached on days 1 of a 21 days cycle. The recommended duration of combination treatment for each patient is at least 8 cycles,
  Other Names: Liposomal doxorubicin hydrochloride

SUMMARY:
Objectives:

Phase I part

* Primary Objective: To determine the recommended dose of the combination of lapatinib with Lipo-Dox as first line chemotherapy in patients with ErbB2 positive metastatic breast cancer.
* Secondary Objectives:To define the safety profile; To observe the response rate and progression free survival

Phase II part

* Primary Objective :To determined the objective response rate of the combination of lapatinib with Lipo-Dox as first line chemotherapy in patients with ErbB2 positive metastatic breast cancer.
* Secondary Objectives:To define the safety profile; To determined the progression free survival

DETAILED DESCRIPTION:
In phase I part Lapatinib (L) - dose level I, II 1000mg po daily dose level III, IV 1250mg po daily Intravenous Lipo Dox at the dose level reached on days 1 of a 21 days cycle• The recommended duration of combination treatment for each patient is at least 8 cycles, then, with continue combination treatment cycles or single lapatinib treatment (start with 1500 mg per day) at investigator's discretion. The treatment will stop if progressive disease, unacceptable toxicity or patient's refusal occurred. Intra patient escalation of dose level is allowed if no major toxicity noted.

In phase II part Patients will receive recommended dose according to phase I study result. The recommended duration of combination treatment for each patient is at least 8 cycles, then, with continue combination treatment cycles or single lapatinib treatment (start with 1500 mg per day) at investigator's discretion. The treatment will stop if progressive disease, unacceptable toxicity or patient's refusal occurred. Intra patient escalation of dose level is allowed if no major toxicity noted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast with evidence of metastatic disease
* Documented ErbB2 over expression or amplified disease in the invasive component of the primary or metastatic lesion as defined by:
* ErbB2 gene amplification by FISH(>6 ErbB2 gene copies per nucleus, or a FISH ratio (ErbB2 gene copies to chromosome 17 signals) of >than 2.2;
* Measurable disease, defined as ≥1 lesion that can be accurately measured in ≥1 dimension as ≥20 mm by conventional techniques OR as ≥10 mm by spiral CT scan
* In phase II part, patients must be chemo-naïve in metastatic setting.
* In phase I part, patient may have received prior chemotherapy in metastatic setting.
* In both phase I and II part, prior Anthracyclines allowed provided total dose of doxorubicin hydrochloride ≤240 mg/m² or epirubicin ≤ 600 mg/m².
* At least 6 months since prior Anthracyclines, and 6 weeks since prior Taxane.
* Patient must be informed and well understand that in current standard of treatment, suggested first line treatments for erbB-2 positive, visceral organ metastatic breast cancer are combination of chemotherapy with herceptin.
* In phase II part, patient must not have exposed to ant-erbB2 targeted therapy treatment in metastatic setting. Herceptin treatment in the neoadjuvant or adjuvant setting is permitted provide that at least 12 months has elapsed since the last dose of herceptin therapy.
* In phase I part, patient may have received prior anti-erbB-2 targeted treatment in metastatic setting.
* Hormone receptor and menopausal status are not specified. Prior treatment with endocrine therapy in the adjuvant or metastatic setting is permitted provided that therapy be discontinued.
* Prior treatments with radiation therapy for palliative management of non-target lesion metastatic disease is permitted provided that at least 2 weeks have elapsed since the last fraction of radiation therapy, disease progression has been documented and all treatment related adverse events are ≦ grade 1 at the time of registration.
* Life expectancy ≥ 12 weeks
* ECOG performance status 0-1
* Patients must have normal organ and marrow function measured within 14 days prior to study entry as defined below:
* WBC ≥ 3,000/mm3
* Absolute neutrophil count ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Normal serum creatinine OR creatinine clearance ≥60 mL/min
* LVEF ≥ 50% (by MUGA)
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow and retain medication
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* Patient consent must be obtained.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Prior therapy with concurrent use of Lapatinib.
* CNS metastasis.
* Ongoing other concurrent investigational agents or anticancer therapy
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious non-healing wound/ulcer/bone fracture, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with GI tract disease resulting in an inability to take medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Phase I part recommended dose of the combination of lapatinib with Lipo-Dox | Phase I: 6 months
  -Phase I part: To determine the recommended dose of the combination of lapatinib with Lipo-Dox

SECONDARY OUTCOMES:
Objective Response Rate | Phase II: 12 months
  -Phase II part: To determined the objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Fang Chiu, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan